CLINICAL TRIAL: NCT02006459
Title: Involvement of Extrapancreatic Factors on Gastrointestinal-mediated Glucose Disposal
Acronym: Px-GIGD
Status: Completed | Type: Observational
Sponsor: University Hospital, Gentofte, Copenhagen (Other)
Collaborators: University of Copenhagen (Other); European Foundation for the Study of Diabetes (Other)
Responsible Party: Principal Investigator, Asger Lund, MD, PhD-student, University Hospital, Gentofte, Copenhagen
Other Study IDs: H-1-2012-123
Record Dates: First submitted 2013-11-27; First posted 2013-12-10 (Estimated); Last update posted 2015-12-02 (Estimated); Status verified 2015-11

CONDITIONS: Diabetes
Keywords: Gastrointestinal-mediated glucose disposal; Total pancreatectomy; Incretin hormones; Glucagon
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — plasma, serum and buffycoat
Oversight: Data Monitoring Committee: No

SUMMARY:
We want to investigate the mechanisms of extrapancreatic effects on gastrointestinal-mediated glucose disposal. In order to do so we will perform oral glucose tolerance tests and isoglycemic intravenous glucose infusions in total pancreatectomised patients and in healthy controls.

DETAILED DESCRIPTION:
In the current project we wish to identify the possible contribution of extrapancreatic effects on gastrointestinal-mediated glucose disposal (GIGD). GIGD reflects the percentage of an individual's glucose disposal following oral glucose tolerance test (OGTT) which is caused by the oral route of glucose administration. In healthy subjects GIGD amounts to ~60%. GIGD describes not only the impact of the incretin effect (insulinotropic substances released upon intestinal stimulation) but includes all factors affecting glucose disposal differently during oral vs. iv administration of glucose (including neural reflexes, activation of afferent nerves in the intestinal mucosa, differences in glucagon secretion, hepatic glucose production and first-pass hepatic uptake of glucose, differences in portal and venous blood glucose concentrations and/or at the present unknown factors. It is likely that the incretin effect (pancreatic effect) constitutes a major contributor to GIGD, but so far it has been impossible to discriminate between pancreatic and extrapancreatic mechanisms underlying GIGD

ELIGIBILITY:
Inclusion Criteria:

* Pancreatectomized patients

  * Caucasians above 18 years of age who have undergone total pancreatectomy
  * Normal haemoglobin
  * Informed consent Healthy Subjects
  * Normal fasting plasma glucose (FPG) and normal HbA1C (according to the World Health Organization (WHO) criteria)
  * Normal haemoglobin
  * Age above 18 years
  * Informed consent

Exclusion Criteria:

* Pancreatectomized patients

  * Inflammatory bowel disease
  * Operation within the last 3 months
  * Ongoing chemotherapy or chemotherapy within the last 3 months
  * Ostomy
  * Nephropathy (serum creatinine >150 µM and/or albuminuria)
  * Severe liver disease (serum alanine aminotransferase (ALAT) and/or serum aspartate aminotransferase (ASAT) >3×normal values)
  * Pregnancy and/or breastfeeding
  * Age above 80 years
  * Any condition that the investigator feels would interfere with trial participation Healthy Subjects
  * Diabetes mellitus (DM)
  * Prediabetes (impaired glucose tolerance and/or impaired FPG)
  * First degree relatives with DM
  * Inflammatory bowel disease
  * Intestinal resection and/or ostomy
  * Nephropathy (serum creatinine >150 µM and/or albuminuria
  * Liver disease (ALAT and/or serum ASAT >2×normal values)
  * Pregnancy and/or breastfeeding
  * Age above 80 years
  * Any condition that the investigator feels would interfere with trial participation

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients operated at/or cared for at the endocrinology out-patient-clinic, Rigshospitalet, University of Copenhagen, Copenhagen Denmark
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2013-09; Primary Completion 2014-09 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Gastrointestinal-mediated glucose disposal (GIGD) | Calculated when the study days are all complete. approximately in 6month
  GIGD will be calculated based on the amounts of glucose utilised during the two glucose administrations forms, OGTT and IIGI (GIGD (%) = 100%×(glucoseOGTT-glucoseIIGI)/glucoseOGTT)
plasma Glucagon | Glucagon will be measured at time points: -30,-15,0,10,20,30,50,70,90,120,150,180 min on all days.

SECONDARY OUTCOMES:
endogenous glucose production | Endogenous glucose production will be calculated based on blood samples at time points: -30,-15,0,10,20,30,50,70,90,120,150,180 min on all days.
  calculated based on infusions of stable isotope marked glucose
Incretin Hormones | incretin hormone levels will be measured at time points: -30,-15,0,10,20,30,50,70,90,120,150,180 min on all days.
  GIP, GLP-1
Satiety, hunger, appetite | Satiety, hunger and appetite will be measured at time points:0,30,60,90,120,150,180 min during each day.
  Will be measured with visual analogue scales (VAS)

CONTACTS AND LOCATIONS:
Locations (1):
- Diabetes Research Division, University Hospital Gentofte, Hellerup, Denmark

REFERENCES:
- [Derived] Lund A, Bagger JI, Wewer Albrechtsen NJ, Christensen M, Grondahl M, Hartmann B, Mathiesen ER, Hansen CP, Storkholm JH, van Hall G, Rehfeld JF, Hornburg D, Meissner F, Mann M, Larsen S, Holst JJ, Vilsboll T, Knop FK. Evidence of Extrapancreatic Glucagon Secretion in Man. Diabetes. 2016 Mar;65(3):585-97. doi: 10.2337/db15-1541. Epub 2015 Dec 15. PMID 26672094